CLINICAL TRIAL: NCT03009149
Title: Effects of Aerobic Exercise on CD4 Count,Viral Load,Selected Psycho-social Trait Among People Living With HIV/AIDS in Nekemte, Ethiopia
Brief Title: Effects of Aerobic Exercise on CD4 Count,Viral Load,Selected Psycho-social Trait
Status: Unknown | Phase: Early Phase 1 | Type: Interventional
Last Known Status: Enrolling by invitation
Sponsor: Mekelle University (Other)
Responsible Party: Principal Investigator, Girma Tilahun, PHD scholar, Mekelle University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Supportive Care
Other Study IDs: ERC0771/2016
Record Dates: First submitted 2016-12-08; First posted 2017-01-04 (Estimated); Last update posted 2017-01-04 (Estimated); Status verified 2016-12

CONDITIONS: HIV
MeSH Terms: interventions — Exercise

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- AEROBIC EXERCISE (Experimental): The effects of 12 week aerobic exercise will record
  Interventions: Other: Aerobic exercise

INTERVENTIONS:
Other: Aerobic exercise — Aerobic exercise will perform 3 days per week

SUMMARY:
H1 - Aerobic exercise will expect to experience significant increase on CD4 counts , reduced viral load , improve psycho-social well being among people living with HIV /AIDS.

DETAILED DESCRIPTION:
Title - Effects of Aerobic Exercise on CD4(cluster of differentiation 4) count , Viral load and Selected Psycho-social Traits Among People Living with HIV/AIDS in Nekemte, Ethiopia

Human being have been challenged with different diseases from time to time. The cause of this diseases are virus , bacteria , fungi and etc. A diseases caused by virus , the Acquired Immune Deficiency Syndrome (AIDS) is very challenging to this century . By the end of 2008, UNAIDS/ world health organization (WHO) estimated that globally, a total of 33.4 million people were living with HIV, where by 31.3 million were adults. In sub-Saharan Africa, 22.4 million people were living with HIV in 2008 . Of these on 15.8 million were under anti-retro viral therapy (ART) to Jun, 2015 and 1.2 mill people died with AIDS related illnesses till end of the 2014 .

Aerobic fitness can improve the health of people living with many diseases, including HIV, and prevents muscle wasting . Exercise benefits may be include cytokine regulation, as is suggested in studies of autoimmune diseases such as multiple sclerosis. Aerobic exercise is one type of rehabilitation strategy that may be used to address disability, such as decreased strength and cardiovascular fitness for persons living with HIV . Exercise may also important to people living with virus because of its link to disease prevention and health promotion. Furthermore, aerobic exercise is creditable of attention because of its connection to body image, which has been shown to be important in certain populations affected by HIV.

This study will conduct in Nekemete town found in east Wollega zone , Oromia regional state. It will be a randomized controlled trial experimental research. The study design will pre-post of experimental clinical trial. Experimental trial will be with intervention of aerobic exercise among people living with HIV/AIDS under ART. The number of sample size is 58. Data analyses will perform with statical analysis for social science (SPSS) version 20. Descriptive data (means, standard deviations (SD) and standard error of the mean (SE), frequency, cross tabulation, charts) will calculate for all variables. The gender difference, viral load, CD4 count, data will analyze using simple t-test and analysis of co-variance (ANCOVA). The level of significance for all analyses will be set at P < 0.05.

ELIGIBILITY:
Inclusion Criteria:

1. Both female and male under ART
2. The distribution of HIV prevalence also varies by age peaking in the 30-40 years age group compared to the other (FDRE,2014) . Because of this the 30-40 will be selected.
3. Participants who have been on first line antiretroviral therapy will be selected.
4. Willing and able to give an informed and agree consent
5. Free of HIV/AIDS related chronic infections that do not allowed aerobic exercise

Exclusion Criteria:

1. Participants with a history of central nervous system dysfunction, hemiparesis (paralysis of one side of the body).
2. Diabetic patients
3. Participant on either as prophylaxis such as the use of antibiotics to prevent infections or as part of (tuberculosis)TB treatment
4. Pregnant and lactating women
5. Free of risk factors those are series cardiac problem
6. Participant who remain in study area throughout the period of study

   -

Ages: 30 Years to 40 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 58 (Estimated)
Dates: Start 2016-11; Primary Completion 2017-01 (Estimated); Study Completion 2017-02 (Estimated)

PRIMARY OUTCOMES:
CD4 count | 12 weeks
  Amount of Cd4 will measure with in one ml blood sample
Effects of aerobic exercise on psycho-social | 12 weeks
  psycho-social will measure by stander questioner called WHOQOL-briff
viral load change duo to aerobic exercise | 12 weeks
  viral load will measured with in one milliliter of blood

CONTACTS AND LOCATIONS:
Overall Officials: Girma Mr Tilahun, MSc, Principal Investigator — phd Scholar

REFERENCES:
- [Background] Terry L, Sprinz E, Stein R, Medeiros NB, Oliveira J, Ribeiro JP. Exercise training in HIV-1-infected individuals with dyslipidemia and lipodystrophy. Med Sci Sports Exerc. 2006 Mar;38(3):411-7. doi: 10.1249/01.mss.0000191347.73848.80. PMID 16540826
- [Background] Terry L, Sprinz E, Ribeiro JP. Moderate and high intensity exercise training in HIV-1 seropositive individuals: a randomized trial. Int J Sports Med. 1999 Feb;20(2):142-6. doi: 10.1055/s-2007-971108. PMID 10190777
- [Background] Stringer WW. HIV and aerobic exercise. Current recommendations. Sports Med. 1999 Dec;28(6):389-95. doi: 10.2165/00007256-199928060-00002. PMID 10623982
- [Background] Smith BA, Neidig JL, Nickel JT, Mitchell GL, Para MF, Fass RJ. Aerobic exercise: effects on parameters related to fatigue, dyspnea, weight and body composition in HIV-infected adults. AIDS. 2001 Apr 13;15(6):693-701. doi: 10.1097/00002030-200104130-00004. PMID 11371683
- [Background] Gomes RD, Borges JP, Lima DB, Farinatti PT. Effects of physical exercise in the perception of life satisfaction and immunological function in HIV-infected patients: Non-randomized clinical trial. Rev Bras Fisioter. 2010 Sep-Oct;14(5):390-5. English, Portuguese. PMID 21180864
- [Background] Ramirez-Marrero FA, Smith BA, Melendez-Brau N, Santana-Bagur JL. Physical and leisure activity, body composition, and life satisfaction in HIV-positive Hispanics in Puerto Rico. J Assoc Nurses AIDS Care. 2004 Jul-Aug;15(4):68-77. doi: 10.1177/1055329003261966. PMID 15296660
- [Background] Perna FM, LaPerriere A, Klimas N, Ironson G, Perry A, Pavone J, Goldstein A, Majors P, Makemson D, Talutto C, Schneiderman N, Fletcher MA, Meijer OG, Koppes L. Cardiopulmonary and CD4 cell changes in response to exercise training in early symptomatic HIV infection. Med Sci Sports Exerc. 1999 Jul;31(7):973-9. doi: 10.1097/00005768-199907000-00009. PMID 10416558
- [Background] O'Brien K, Nixon S, Tynan AM, Glazier R. Aerobic exercise interventions for adults living with HIV/AIDS. Cochrane Database Syst Rev. 2010 Aug 4;2010(8):CD001796. doi: 10.1002/14651858.CD001796.pub3. PMID 20687068
- [Background] Nixon S, O'Brien K, Glazier RH, Tynan AM. Aerobic exercise interventions for adults living with HIV/AIDS. Cochrane Database Syst Rev. 2005 Apr 18;(2):CD001796. doi: 10.1002/14651858.CD001796.pub2. PMID 15846623
- [Background] Nixon S, O'Brien K, Glazier RH, Tynan AM. Aerobic exercise interventions for adults living with HIV/AIDS. Cochrane Database Syst Rev. 2002;(2):CD001796. doi: 10.1002/14651858.CD001796. PMID 12076422